CLINICAL TRIAL: NCT04331197
Title: Effect of High BMI on Ovulation Induction Using Letrozole Versus Clomid
Brief Title: BMI Effect on the Response to Ovulation Induction in Letrozole vs Clomid
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Elkattan, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol 600
Record Dates: First submitted 2020-03-27; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Subfertility
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Letrozole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clomiphene Citrate-High BMI women (Active Comparator): Clomid 50 mg, 2 tablets orally every day from day 2-5 of the period for 5 days
  Interventions: Drug: Clomiphene Citrate 50mg
- Letrozole-High BMI women (Active Comparator): Femara 2.5 mg, 2 tablets orally every day from day 2-5 of the period for 5 days
  Interventions: Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: Clomiphene Citrate 50mg — Clomid 50 mg, 2 tablets orally every day from day 2-5 of the period for 5 days
  Other Names: Clomid
  Arms: Clomiphene Citrate-High BMI women
Drug: Letrozole 2.5mg — Femara 2.5 mg, 2 tablets orally every day from day 2-5 of the period for 5 days
  Arms: Letrozole-High BMI women

SUMMARY:
There is an increased prevalence of high Body mass index (BMI) all over the world.High BMI is shown to have an impact on the female reproductive system.It can contribute to both ovulatory and anovulatory subfertility.

Clomiphene citrate and Letrozole have been used for treatment of infertility.Both are used for induction of ovulation.

Clomiphene citrate is an estrogen receptor antagonist .It increases serum FSH and it has its limitation due to his antiestrogenic effect,it has an ovulation rate 70-80% but pregnancy rate is only 22% because of its anti-estrogenic effect on endometrium and poor cervical mucus (Legro RS et al.,2007) Letrozole is an aromatase inhibitor which inhibits the production of estrogen, which influences the action of the brain's hypothalamus and pituitary on the functioning of the ovaries by increasing FSH.Due to the antiestrogenic effect of clomiphene citrate,Letrozole can be used as an alternative.

The investigators are comparing the effect of both medications on the outcome of the induction of ovulation in women with high BMI.

DETAILED DESCRIPTION:
This is a Randomized controlled trial .The researchers include160 women with BMI more than 30 who were suffering from subfertility for more than 2 years. The investigators will randomise them into 2 groups. Group A:They were prescribed 100 mg of clomiphene citrate from day 2-5 of the cycle for 5 days. Group B : They were prescribed 5 mg of Letrozole from day 2-5 of the cycle.

Vaginal ultrasound was performed on day 11 of the cycle, After at least one follicle reached 15 mm, The patient was encouraged to have sexual intercourse every other day for few days.The patients will have a midluteal progesterone level to confirm ovulation and will have a pregnancy test in 2 weeks if missed period. The researchers will compare the number of mature follicles, endometrial thickness on the day when there are mature follicles, occurrence of pregnancy, multiple pregnancies, and miscarriages .

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years old.
* History of subfertility for 2 years.
* No previous IVF
* Intact tubes as evidenced by HSG or Hycosy
* Normal Sperm parameters according to WHO criteria.
* Ability to have regular intercourse during the ovulation induction phase of the study.

Exclusion Criteria:

* Age less than 18 years old or older than 45 years old.
* FSH> 15 mIU/ml
* Tubal factor of infertility
* Male factor of infertility
* Current pregnancy,abnormal uterine bleeding.
* History of use of hormonal contraception in the last 3 months.
* Untreated medical problems: thyroid disease,hyperprolactinemia or contraindication to pregnancy as uncontrolled diabetes or severe heart disease.
* Contraindications to clomiphene citrate: hypersensitivity to clomid.
* Contraindications to letrozole: hypersensitivity to letrozole .

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of ovulation | day 21 of 28 day cycle or 7 days post LH surge
  Raised concentration of serum progesterone

SECONDARY OUTCOMES:
Number of mature follicles | day 12-19 of the cycle (At the end of the treatment cycles, each cycle 28 days)
  Number of follicles> 15mm
Endometrial thickness | day 12-19 of the cycle (At the end of the treatment cycles, each cycle 28 days)
  the thickest part of the endometrial lining at the longitudinal plane at the time of mature follicle
Conception | 4-5 weeks post treatment
  Number of participants with positive pregnancy test (serum or urine),serum BHCG > 25 IU/L
clinical pregnancy | 6 weeks post treatment
  Number of participants with gestational sac with positive fatal pulsation

IPD SHARING:
Plan to Share IPD: Undecided